CLINICAL TRIAL: NCT04575220
Title: Pilot Study of Adaptive Home Based Pulmonary Tele-exercise (AHTE)
Brief Title: Adaptive Home Based Pulmonary Tele-exercise
Acronym: AHTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh Ann Callahan, MD (Other)
Responsible Party: Sponsor-Investigator, Leigh Ann Callahan, MD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58756
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Rehabilitation

STUDY DESIGN:
Intervention Model Description: Single arm pilot study evaluating fitness before and after home based rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tele-exercise (Experimental): Subjects will perform three sessions/week of home exercise using bicycles for 12 weeks
  Interventions: Other: 12 weeks of bicycle exercise

INTERVENTIONS:
Other: 12 weeks of bicycle exercise — Subjects will conduct monitored exercise, three sessions per week for 12 weeks.

SUMMARY:
The goal of this pilot study is to determine if a home based bicycle exercise program can significantly improve the exercise tolerance and well being of pulmonary outpatients. The investigators will use a computer based monitoring system to allow us to speak with participants, view participants, and track patient bicycle activity (speed, duration of exercise, rate of work) during exercise sessions. The investigators plan to have participants perform three telemonitored exercise sessions per week for 12 weeks as part of this program. The investigators will assess exercise performance on the bicycle, called a work rate test, at the beginning of the program and then again at 6 weeks and 12 weeks into the program to determine if the program can produce a clinically significant improvement in work rate test performance (i.e. a greater than 1.15 minute increase in exercise duration at an 80% work rate). The investigators will also assess participant CRQ, SPPB scores and SF36 scores (indices of patient well being) at baseline, at 6 weeks, and at 12 weeks, to determine if the exercise program elicits an increase in these indices.

DETAILED DESCRIPTION:
Studies have shown that pulmonary rehabilitation, which includes exercise and patient education, is a valuable therapy for patients with pulmonary diseases. In fact, pulmonary rehabilitation delivered soon after patient discharge is known to produce a major improvement in patient outcomes. Specifically, studies have shown this intervention reduces readmission rates by 30-70% over the next year. In addition, this therapy improves exercise tolerance, performance of tasks of daily living and sense of patient well being. One study even shows this therapy is 30 times as effective as bronchodilator therapy in improving patient outcomes.

Surprisingly, however, very few pulmonary patients receive pulmonary rehabilitation. Recent studies have shown that 94-98% of discharged pulmonary patients fail to receive this therapy. This pattern has been shown to exist across the United States, with no state demonstrating a much larger use of this therapy. Moreover, use of this therapy is even worse for minorities (only 1% receive pulmonary rehabilitation) and rural populations, such as patients in southern and eastern Kentucky. Several factors are responsible for this failure to employ pulmonary rehabilitation including: (a) very few centers are available and patients cannot realistically travel to the existing centers because of distance, (b) this form of rehabilitation is expensive and patients must pay a large copay (30-50 dollars per session, adding up to a total of 1800 dollars for a typical 12 week program) which many patients cannot afford, (c) centers are only open for restricted hours and working patients cannot miss work to go for rehabilitation, and (d) patients are only eligible for 36 treatment sessions for life.

The purpose of the present project is to define a new home based exercise program that should provide exercise training as good or better than conventional brick and mortar rehabilitation programs. The investigators will use technological advances in home based exercise equipment to both precisely measure participant exercise and to assess physiological improvements over time. This technology will also reduce the expense required to supervise participant training, dramatically reducing costs compared to conventional center based programs. In addition, because programs are home based, the investigators can provide access to participants in rural locations, reduce travel, and easily extend the convenience and schedule of training sessions to accommodate participant lifestyles. While recently there have been a few attempts to provide home based pulmonary rehabilitation programs (e.g. by VA rural health, the Southern Alabama consortium) these other programs do not provide the intensity of training possible with the new paradigm in the current project, are not proven to have the same beneficial effects as conventional center based rehabilitation, and have higher personnel costs making long term financial viability uncertain.

ELIGIBILITY:
Inclusion Criteria

* age from 18-80 years
* previous diagnosis of pulmonary disease, including known chronic pulmonary diseases (COPD, ILD), recent admission for pulmonary disease (pneumonia, asthma, obstructive lung disease), recent ICU discharge for a diagnosis of respiratory failure, and/or previous COVID-19 disease with demonstration of recovery (two negative antigen tests)
* the capacity to perform cycling exercise

Exclusion Criteria

* if the physician caring for the patient determines that the patient should not participate in a home based exercise program
* if the patient has active ischemic cardiac disease
* if the patient's home does not have sufficient space or internet connectivity for the computer and bicycle to be operative
* if the patient is a pregnant female
* if the patient is a prisoner
* if the patient is institutionalized
* if the patient has a terminal clinical condition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
80% work rate test | This will be measured at baseline, at 6 weeks, and at 12 weeks. The primary outcome measure to be assessed is the change in the 80% work rate test time between the initial and 12 week assessment.
  This will measure changes in the time the subject can exercise at 80% of the maximum work rate.

SECONDARY OUTCOMES:
CRQ score: Chronic Respiratory Questionnaire | baseline and at 6 weeks and 12 weeks
  this will ask how short of breath the subject is: Scores will range from 20 to 140, the higher the score, the better the patient's condition
SF36: Short Form Survey; 36 Questions | baseline and at 6 weeks and 12 weeks
  this questionnaire will ask about quality of life; each question scores from 1 to 6; the higher the score, the worse the patients' condition
SPPB: Short Physical Performance Battery | baseline and at 6 weeks and 12 weeks
  this will test the ability to perform simple movements; balance will be scores 0 to 4, gait speed 2 to 8, and chair standing 0 to 4; the higher the score, the better the patient's condition

CONTACTS AND LOCATIONS:
Locations (1):
- Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No